CLINICAL TRIAL: NCT01243983
Title: A Multi-Center, Double-Masked, Parallel-Group, Placebo-Controlled Study to Assess the Efficacy and Safety of Voclosporin as Therapy in Subjects With Active Noninfectious Uveitis Involving the Intermediate and/or Posterior Segments of the Eye
Brief Title: Efficacy and Safety of Voclosporin to Treat Active Noninfectious Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lux Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX211-11; 2010-022128-63 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Noninfectious Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LX211 (Experimental)
  Interventions: Drug: LX211
- Placebo (Placebo Comparator)
  Interventions: Drug: LX211

INTERVENTIONS:
Drug: LX211 — Subjects will be sequentially assigned to one of the following treatment arms in a 1:1 ratio:
  * Treatment Arm A: voclosporin 0.4 mg/kg p.o. b.i.d., not to exceed 40 mg p.o. b.i.d.
  * Treatment Arm B: placebo p.o. b.i.d.
  Dosage Form:
  • Soft gelatin capsule
  Duration of treatment:
  • 24 weeks

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of voclosporin as therapy in subjects with active noninfectious uveitis involving the intermediate and/or posterior segments of the eye (i.e., anterior + intermediate-, intermediate-, posterior- or pan-uveitis).

ELIGIBILITY:
Inclusion Criteria:

* Active noninfectious uveitis involving the intermediate and/or posterior segment (i.e., anterior + intermediate-, intermediate-, posterior- or pan-uveitis) in at least one eye as evidenced by a vitreous haze grade of at least 2+ at the baseline visit. Subjects who also have anterior segment involvement need not be excluded if otherwise qualified.
* Subjects must be:

  * Capable of understanding the purpose and risks of the study.
  * Able to give written informed consent.
  * Able to comply with all study requirements.

Exclusion Criteria:

* Ocular Disease/Conditions
* The following conditions are exclusionary if present:

  * Uveitis limited to only the anterior segment of the study eye.
  * Confirmed or suspected infectious uveitis in either eye.
* Prior and Current Treatment:

  - As defined in the protocol
* Extraocular Conditions:

  - As defined in the protocol.
* Laboratory, Blood Pressure and ECG Evaluations:

  * As defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The change from baseline in graded vitreous haze in the study eye at 12 weeks of therapy or at the time of treatment failure, if earlier. | 12 weeks

SECONDARY OUTCOMES:
Daily mean systemic corticosteroid dose used during Weeks 12-24 | Weeks 12-24
Time to augmentation with corticosteroid therapy. | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Anglade, M.D., Study Chair — Chief Medical Officer
Locations (49):
- United States (27):
  - Peoria, Arizona
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Mountain View, California
  - Sacramento, California
  - Santa Ana, California
  - Torrance, California
  - Indianapolis, Indiana
  - Ellsworth, Maine
  - Baltimore, Maryland
  - Cambridge, Massachusetts
  - Newark, New Jersey
  - Belmont, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Dublin, Ohio
  - Middleburg Heights, Ohio
  - Ashland, Oregon
  - Philadelphia, Pennsylvania
  - Ladson, South Carolina
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
- Vienna, Austria
- Brazil (3):
  - Recife
  - Rio de Janeiro
  - São Paulo
- Ottawa, Ontario, Canada
- Czechia (4):
  - Brno
  - Hradec Králové
  - Olomouc
  - Prague
- France (3):
  - Angers
  - Bordeaux
  - Paris
- Germany (2):
  - Münster
  - Tübingen
- Italy (5):
  - Bologna
  - Milan
  - Padua
  - Parma
  - Reggio Emilia
- United Kingdom (3):
  - Birmingham
  - London
  - York